CLINICAL TRIAL: NCT05492994
Title: Longitudinal Study Without an Investigational Medicinal Product in Patients With Progressive Fibrosing Interstitial Lung Disease (PF-ILD) to Evaluate Novel Imaging-based Biomarkers in Comparison With Lung Function for Use in Early Clinical Development
Brief Title: A Study to Test Different Imaging Techniques in Patients With Different Types of Interstitial Lung Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0352-2157
Record Dates: First submitted 2022-08-08; First posted 2022-08-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Spirometry; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Progressive Fibrosing Interstitial Lung Disease (PF-ILD) (Experimental)
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO); Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Chest Computer Tomography; Diagnostic Test: Blood biomarker analysis

INTERVENTIONS:
Diagnostic Test: Spirometry — Pulmonary function test
Diagnostic Test: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) — Pulmonary function test
Diagnostic Test: Magnetic Resonance Imaging — Magnetic Resonance Imaging
Diagnostic Test: Chest Computer Tomography — Chest Computer Tomography
Diagnostic Test: Blood biomarker analysis — Blood biomarker analysis

SUMMARY:
The main objectives of this imaging biomarker study are to assess the annual lung function change in patients with progressive fibrosing interstitial lung disease (PF-ILD) including idiopathic pulmonary fibrosis (IPF), with Usual Interstitial Pneumonia (UIP) or probable UIP Computer Tomography (CT) pattern, and to monitor lung structural changes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the study.
2. Patients with a documented diagnosis of Progressive Fibrosing Interstitial Lung Disease (PF-ILD) including Idiopathic Pulmonary Fibrosis (IPF), with Usual Interstitial Pneumonia (UIP) or probable UIP chest Computer Tomography (CT) pattern and no anti-fibrotic treatment (nintedanib or pirfenidone) at baseline and previously (treatment-naive regarding Standard of Care (SoC))
3. Male or female patients aged ≥ 40 years when signing the informed consent.
4. Forced Vital Capacity (FVC) ≥ 45% predicted of normal reviewed at Visit 1.
5. Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) corrected for Haemoglobin ≥ 25% of predicted normal reviewed at Visit 1.
6. Body mass index (BMI) <=30 kg/m2 reviewed at Visit 1.
7. Glomerular filtration rate (GFR) ≥30 ml/min reviewed at Visit 1.
8. Supportive Thyroid-Stimulating Hormone (TSH) evaluation for all participants >60 years and/or history of thyroid disease according to local standard procedures at Visit 1.

Exclusion Criteria:

1. Significant pulmonary disease other than PF-ILD or other medical conditions (as determined by medical history, examination and clinical investigations at screening) that may, in the opinion of the investigator result in any of the following:

   * Put the patient at risk because of participation in the study
   * Influence the results of the study
   * Cause concern regarding the patient's ability to participate in the study Patients with a history of a documented Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection will be excluded if lung changes due to the infection have been observed at screening (on discretion of the investigator).
2. Any documented active or suspected malignancy or history of malignancy on discretion of the investigator.
3. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the accurate assessment of endpoints of the study.
4. Patients not able to understand or follow study procedures or patients not expected to comply with the protocol requirements or not expected to complete the study as scheduled (e.g., chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable study participant).
5. Previous enrolment in this study.
6. Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s) or receiving other investigational treatment(s).
7. Women who are pregnant, nursing, or who plan to become pregnant while in the study. Women of childbearing potential1 not willing or able to use highly effective methods of birth control per International Council for Harmonisation (ICH) M3 (R2). A list of contraception methods meeting these criteria is provided in the patient information and in the study protocol.
8. Life expectancy for disease other than Interstitial Lung Disease (ILD) <2.5 years (investigator assessment) Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Absolute change in Forced Vital Capacity (FVC) % predicted from baseline to week 52 | at baseline and at week 52

SECONDARY OUTCOMES:
Absolute change in fibrosis extent in % of lung volume determined on chest Computer Tomography (CT) from baseline to week 52 | at baseline and at week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com
- See also: Related Info — https://mhh-jvc.de/team